CLINICAL TRIAL: NCT05623839
Title: A Multiple Dose Titration Study in Participants With Obesity or Overweight to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3305677
Brief Title: A Study of LY3305677 in Participants With Obesity Or Overweight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18522; I8P-MC-OXAG (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-11-15; First posted 2022-11-21 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3305677 (Experimental): LY3305677 administered subcutaneously (SC)
  Interventions: Drug: LY3305677
- Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3305677 — Administered SC
  Arms: LY3305677
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn about the safety and tolerability of LY3305677 when given to participants with obesity or overweight. Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body. Each enrolled participant will receive injections of LY3305677 or placebo given just under the skin. For each participant, the study will last about approximately 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation
* Participants with stable weight for 3 months and body mass index of 27.0 and 50.0 kilograms per square meter (kg/m²)

Exclusion Criteria:

* Have history of type 1 diabetes mellitus or type 2 diabetes mellitus, ketoacidosis, or hyperosmolar state or coma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Week 20
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3305677 | Predose up to 72 hours postdose
  PK: Cmax of LY3305677
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3305677 | Predose up to 72 hours postdose
  PK: AUC of LY3305677
Pharmacodynamics (PD): Percentage change in Body Weight | Baseline through Week 20
  PD: Percentage change in Body Weight

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - ICON Early Phase Services, San Antonio, Texas
  - ICON Early Phase Services Lenexa Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhattachar SN, Tham LS, Li Y, Chua L, Ng SX, Tang Y, Ibriga H, Ni W, Gurbuz S, Mather KJ, Thomas MK. Mazdutide reduces body weight in adults with overweight or obesity: A high-dose Phase 1 trial. Diabetes Obes Metab. 2025 Nov;27(11):6460-6469. doi: 10.1111/dom.70040. Epub 2025 Aug 20. PMID 40832785